CLINICAL TRIAL: NCT02133157
Title: Phase I Study of Safety and Pharmacokinetics of Sulfatinib(HMPL-012) in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of Sulfatinib(HMPL-012) in Patients With Advanced Solid Tumors
Acronym: HMPL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-012-00CH1
Record Dates: First submitted 2014-03-08; First posted 2014-05-07 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Tumor
Keywords: tumor
MeSH Terms: conditions — Neoplasms | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulfatinib capsule (Experimental): cohort 1: Sulfatinib single oral dosing;after 7days,Sulfatinib continuous oral dosing ( once a day) 28days as a cycle.
  Interventions: Drug: Sulfatinib

INTERVENTIONS:
Drug: Sulfatinib — Sulfatinib is a capsule in the form of25, 50mg , 100mg; oral, once a day
  Other Names: HMPL-012

SUMMARY:
Sulfatinib (HMPL-012) is a novel oral small molecule that selectively inhibits vascular endothelial growth factor receptors (VEGFR) 1, 2, and 3 and inhibits FGFR kinase activity has demonstrated potent inhibitory effects on multiple human tumor xenografts. This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and recommended dose for phase II ,to evaluate the pharmacokinetics , safety and preliminary anti-tumor activity of HMPL-012 at single doses and multiple doses .

DETAILED DESCRIPTION:
This will be an open-label, phase I study. This study will evaluate the safety and pharmacokinetics of HMPL-012 after a single administration followed by a 28-Day continuous course of therapy; evaluate the safety and preliminary efficacy in an open-label administration of at the MTD. All subjects of this study will be permitted to continue therapy with only safety monitoring and monthly assessments for progression, if the product is well tolerated and the subject has stable disease or better

ELIGIBILITY:
Inclusion Criteria:

•≥ 18 and ≤ 70 years of age

* Histological or cytological confirmed solid malignant tumor
* ECOG performance status of 0-2
* Standard regimen failed or no standard regimen available
* Life expectancy of more than 12 weeks
* LVEF ≥ 50%

Exclusion Criteria:

* Pregnant or lactating women
* Adequate hepatic, renal, heart, and hematologic functions (platelets <75 × 109/L, neutrophil <1.5 × 109/L, hemoglobin < 90g/dl ,serum creatinine within upper limit of normal(ULN), total bilirubin and serum transaminase within upper limit of normal(ULN), and PT, APTT, TT, Fbg normal
* Any factors that influence the usage of oral administration
* Evidence of uncontrolled CNS metastasis
* Intercurrence with one of the following: non-controlled hypertension, coronary artery disease, arrhythmia and heart failure
* Abuse of alcohol or drugs
* Less than 4 weeks from the last clinical trial
* Previous treatment with VEGF/VEGFR inhibition
* Disability of serious uncontrolled intercurrence infection
* Uncontrolled hemorrhage in GI
* Within 12 months before the first treatment occurs artery/venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack) etc.
* Within 6 months before the first treatment occurs acute myocardial infarction, acute coronary syndrome or CABG
* Bone fracture or wounds that was not cured for a long time
* Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To assess number of participants with adverse events as a measure of safety and tolerability during dose escalating | 1-28days after every drug administration
  The primary endpoint is evaluation of safety during the first 28-day cycle 1 of therapy following the initiation of multiple dosing of HMPL-012. The safety variables to be evaluated in this study are adverse events, physical examinations, vital signs (specifically including blood pressure), clinical laboratory evaluations including serum chemistry, hematology , and urinalysis (with detailed sediment analysis, proteinuria, and 24-hour urine for collection for protein), and electrocardiograms (ECGs) in triplicate

SECONDARY OUTCOMES:
To measure the plasma concentration of HMPL-012 in single and repeated doses | Day 1-3 Single Dose and Day 1-56 Steady State
  In the study of single-dose, full PK profiles of HMPL-012 will be obtained following administration of a single oral dose of HMPL-012 on Day 1 to Day 3. At multiple-dose, PK sampling will include a pre-dose and at the 1,4,8,12 hour time points on days 1,14,28 of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2, 3, 7, 15 and 29 of the first 28-Day cycle of therapy and pre-dose on days 56 of the cycle 2.

OTHER OUTCOMES:
Objective Response Rate | every 4 weeks until 1 year
  Anti-tumoral efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors (RECIST v 1.0) at baseline (Day -14 to -1) and at the end of two 28-Day cycles of therapy . For patients that continue on repeat 28-Day cycles after the primary evaluation period, progression will be assessed after each two 28-Day cycles of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ming J Xu, PHD, Principal Investigator — Academy of Military Medical Affiliated Hopital
Locations (1):
- Academy of Military Medical Affiliated Hopital, Beijing, China